CLINICAL TRIAL: NCT05701605
Title: Prognostic and Diagnostic Roles of Some Non-classic Biomarkers in Pediatric Pneumonia
Brief Title: Roles of Some Non-classic Biomarkers in Pediatric Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nahla Sameh Abd El-Aleem Mahmoud, Principal Investigator, Assiut University
Other Study IDs: Pneumonia biomarkers
Record Dates: First submitted 2022-12-17; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Pneumonia in Children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The current work aims to:

1. Measure the levels of Neutrophil CD64 Receptor, Monocyte Human Leukocyte Antigen-DR (mHLA-DR), and Triggering Receptor Expressed on Myeloid Cells 1 (TREM-1) in children suffering from pneumonia.
2. Compare these levels to their levels in healthy control children.
3. Analyze the cut-off point, sensitivity, specificity, and area under the ROC curve of these biomarkers to test their abilities to early differentiate children with pneumonia from healthy control children.
4. Conclude or reject their possible use as diagnostic and/or prognostic markers in pediatric pneumonia.

DETAILED DESCRIPTION:
Pneumonia is the world's leading infectious cause of mortality. It is one of the most common lower respiratory tract infections, which contributes significantly to the burden of antibiotic use. Because of the complexity of the pathophysiology, pneumonia is widely recognized that the clinical diagnosis and prognosis are usually not enough to accurately estimate the severity of the condition. The most difficult task for a doctor is above all the value of risk in patients with community-acquired pneumonia. Early diagnosis is important to reduce hospitalization and death.

There are widespread biomarkers, none of which looks perfect, and the demand for new biomarkers that maximizes the severity and treatment response for pneumonia has increased. Indirect methods are utilized to isolate the organism. These include polymerase chain reaction of throat swab, gram stain, culture of nasopharyngeal aspirate, and blood cultures. However, interpretation can be difficult as children are found to be asymptomatic carriers of a range of organisms and a positive result on PCR may not be indicative of the cause of CAP. C-reactive protein, and White blood cell count are often part of the diagnostic workup in an inpatient setting. However, the changes observed are not specific to predict causative pathogens. Instrumental diagnostics, such as a chest X-ray are not sensitive or specific and are not recommended in the initial diagnosis of a suspected community acquired pneumonia.

Biomarkers in pneumonia may be the ones that indicate inflammation or may be released specifically, after lung injury due to infection. The measured levels of biomarkers should be interpreted cautiously and always be correlated with clinical findings as many confounding factors should be taken into consideration for interpretation. Factors like age, antibiotic pretreatment, chronic hepatic disease, corticosteroids, renal impairment, and viral confection can critically affect some biomarker levels and thus their sensitivity and specificity regarding treatment failure and clinical stability. Hence, results should be interpreted in line with the clinical presentation, and they should never substitute clinical judgment.

The importance of the classic biomarkers such as procalcitonin and C-reactive protein has been declined. The limitations of PCT are being elevated in a variety of noninfectious conditions, such as cirrhosis, pancreatitis, mesenteric infarction, burns, and aspiration pneumonitis. Also, its diagnostic and predictive value declines in patients with severe sepsis and in localized infections (e.g., endocarditis, empyema). Studies differ as to what are the appropriate negative cut-off points for PCT. Criticism of the role of CRP in diagnostics includes not only the delay in response to clinical stimulus but also its poor specificity as it is elevated in a variety of pathologies, such as trauma, surgery, burns, and immunological-mediated inflammatory diseases. Mendez et al. successfully demonstrated that CRP is a significant independent predictor for the absence of severe complications in CAP.

The establishment of new biomarkers in clinical practice would not only facilitate accurate diagnosis but would also help to reduce the amount of antibiotics used. Burgos etal. [2016] assess the usefulness of neutrophil CD64 expression to identify patients with community-acquired pneumonia (CAP) at risk of a poor outcome. The sensitivity/specificity of nCD64 in predicting poor outcome [defined as intensive care unit (ICU) admission and/or clinical deterioration after arrival at the emergency department] was calculated. Although nCD64 expression is associated with an increased risk of ICU admission or clinical deterioration after admission, its accuracy in predicting these poor outcomes is modest and does not significantly improve the predictive ability of severity scores. Qun and Mei-Yu [2012], studied the clinical value of the expression of neutrophil surface CD64 in the diagnosis of community-acquired pneumonia in children. They found that ROC curve analysis showed that the threshold of CD64 and CRP was 2.8 and 8 mg/L respectively. Specificity of CD64 index (90%) was much higher than CRP (74%). They stated that the determination of peripheral blood neutrophil CD64 contributes to the early diagnosis of pulmonary bacterial infection and the evaluation of the anti-infection effect.

Zhuang etal., [2015] study the level of monocyte-human leukocyte antigen-DR (mHLA-DR), an immune function-related biomarker, at 24 h after admission, to predict the outcomes of subjects with severe pneumonia. They found that mHLA-DR may be a reliable biomarker that can predict the outcomes of patients with severe community-acquired pneumonia, and 27.2% may be the cut-off value to predict the outcomes. They reported that non-survivors significantly expressed reduced levels of mHLA-DR on their monocyte membranes. There is still not enough evidence whether mHLA-DR could be a useful marker in CAP.

Triggering receptor expressed on myeloid cells 1 (TREM-1) is an inflammatory receptor that causes inflammation after exposure to extracellular fungi and bacterial pathogens. Elevated TREM-1 levels are a potential marker of lung disease. El Nady etal. [2019] found that TREM-1 level was significantly higher in ventilated children with pneumonia compared to the control group (1). Grover et al. [2014] found that TREM-1 is a good predictor of ventilator-associated pneumonia (VAP) ; however, Palazzo et al. 2012 claimed that TREM-1 can be found elevated in the bronchoalveolar lavage (BAL) fluid of patients with and without confirmed VAP. Therefore, further studies are required to fully determine the diagnostic power of TREM-1 for VAP.

ELIGIBILITY:
Inclusion Criteria:

1. Children more than one month and till age of 5 years
2. Clinical diagnosis of CAP.

Exclusion Criteria:

1) All pediatric patients with comorbidities and diagnosed with CAP as: severe sepsis& localized infections e.g., endocarditis, empyema& autoimmune diseases& liver cirrhosis& children receiving immunosuppressive therapy.

Ages: 1 Month to 5 Years | Sex: All
Age Groups: Child
Study Population: 60 infant and child aged 1 month to 5 years with pneumonia and 60 normal infant and child of comparable age and sex as control.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Measure the level of Neutrophil CD64 Receptor | Baseline
  a peripheral blood neutrophil CD64
Measure the level of Monocyte Human Leukocyte Antigen-DR (mHLA-DR) | Baseline
  an immune function-related biomarker
Measure the level of Triggering Receptor Expressed on Myeloid Cells 1 (TREM-1) | Baseline
  an inflammatory receptor that causes inflammation after exposure to extracellular fungi and bacterial pathogens

CONTACTS AND LOCATIONS:
Overall Officials: El-Sayed Khalil, Prof, Principal Investigator — Assiut University; Yasser Farouk, Assist prof, Principal Investigator — Assiut University; Khalid Mohany, Assist prof, Principal Investigator — Assiut University